CLINICAL TRIAL: NCT02338349
Title: A Phase I, Multicenter, Open-Label, Multi-Part, Dose-escalation Study of RAD1901 in Postmenopausal Women With Advanced Estrogen Receptor Positive and HER2-Negative Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAD1901-005
Record Dates: First submitted 2014-12-31; First posted 2015-01-14 (Estimated); Last update posted 2022-08-18 (Actual); Status verified 2020-05

CONDITIONS: Advanced ER+, HER2-Negative Breast Cancer
MeSH Terms: interventions — elacestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elacestrant (Experimental): Part A, Dose Escalation: Patients will be assigned sequentially to escalating doses of elacestrant.
  Part B, Safety Expansion: Once the MTD has been identified and/or a RP2D has been selected, additional patients will be enrolled to further evaluate the safety, tolerability and preliminary efficacy of the RP2D.
  Part C, Tablet Introduction: A cohort of patients will be enrolled to evaluate the safety, tolerability, and PK of a tablet dosage form at 400 mg QD.
  Part D, Dose Expansion: A cohort of patients will be enrolled to evaluate the safety, tolerability, PK and preliminary anti-tumor effect of elacestrant in tablet dosage form at 400 mg QD PO in a group of patients with a more homogeneous prior treatment history
  Interventions: Drug: Elacestrant

INTERVENTIONS:
Drug: Elacestrant

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and preliminary efficacy of elacestrant (RAD1901) in patients with advanced ER+, HER2-negative breast cancer.

DETAILED DESCRIPTION:
The primary objective is to determine the maximum tolerated dose (MTD) and/or recommended Phase 2 dose (RP2D) of elacestrant in patients with advanced ER+HER2-negative breast cancer.

The secondary objectives of this study are:

* To assess the safety and tolerability of elacestrant
* To evaluate the pharmacokinetics (PK) of elacestrant
* To evaluate the preliminary anti-tumor effect of elacestrant

ELIGIBILITY:
Key Inclusion Criteria:

1. Patients must be post-menopausal women, as defined in the protocol
2. 18 years or older
3. Patients with histological or cytological proven diagnosis of adenocarcinoma of the breast with evidence of either locally advanced, inoperable and/or metastatic disease
4. Part A, B, C: Patients must have received no more than 2 prior chemotherapeutic regimens and at least 6 months of prior endocrine therapy
5. Part D: Patients may have received up to 1 previous line of chemotherapy and must have previously received 2 or more lines of endocrine therapy for advanced/metastatic breast cancer as a single agent or in combination. Patients must have received fulvestrant as one of the previous lines of endocrine therapy and have had documented progression while on, or within 1 month after the end of, fulvestrant therapy for advanced/metastatic breast cancer. Patients must have received prior treatment with a CDK4/6 inhibitor

Note: This list is not complete. Further inclusion criteria is provided in the protocol synopsis.

Key Exclusion Criteria:

1. Prior anticancer or investigational drug treatment within the following windows:

   1. Tamoxifen therapy less than 14 days before first dose of study treatment
   2. Part A, B and C: Fulvestrant therapy less than 90 days before first dose of study treatment. Part D: Fulvestrant therapy less than 42 days before first dose of study treatment
   3. Any other anti-cancer endocrine therapy less than 14 days before first dose of study treatment
   4. Any chemotherapy less than 28 days before first dose of study
   5. Any investigational drug therapy less than 28 days or 3 half-lives (whichever is longer) prior to first dose of study treatment
2. Patients with untreated or symptomatic central nervous system (CNS) metastases
3. Patients with endometrial disorders, including evidence of endometrial hyperplasia, dysfunctional uterine bleeding or cysts

Note: This list is not complete. Further exclusion criteria is provided in the protocol synopsis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | The first 28 days of treatment.
  To determine the maximum tolerated dose (MTD) and/or recommended Phase II dose (RP2D) of Elacestrant (RAD1901), the incidence of Dose Limiting toxicities (DLTs) will be assessed.

SECONDARY OUTCOMES:
Safety and Tolerability of Elacestrant (RAD1901) | Up to 30 days after the end of treatment.
  Safety and tolerability will be assessed in terms of adverse events, serious adverse events, ECG, physical examination, vital signs, and laboratory values.
Pharmacokinetics of Elacestrant (RAD1901) | Every 28 days
  Plasma concentrations of RAD1901 will be assessed at predefined intervals
Anti-Tumor Effect of Elacestrant (RAD1901) | Every 8 weeks
  Tumor response will be evaluated in patients with measurable or evaluable disease, using RECISTv1.1 guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Director, Clinical Operations, Study Director — Radius Pharmaceticals, Inc
Locations (1):
- Radius Pharmaceuticals, Inc., Waltham, Massachusetts, United States

REFERENCES:
- [Derived] Bardia A, Kaklamani V, Wilks S, Weise A, Richards D, Harb W, Osborne C, Wesolowski R, Karuturi M, Conkling P, Bagley RG, Wang Y, Conlan MG, Kabos P. Phase I Study of Elacestrant (RAD1901), a Novel Selective Estrogen Receptor Degrader, in ER-Positive, HER2-Negative Advanced Breast Cancer. J Clin Oncol. 2021 Apr 20;39(12):1360-1370. doi: 10.1200/JCO.20.02272. Epub 2021 Jan 29. PMID 33513026